CLINICAL TRIAL: NCT06023524
Title: The Effectiveness Combination of Laser Acupuncture and Standard Medication on Pain Score, Interincisal Distance and Swelling in Mandibular Third Molar Post-Odontectomy Patients
Brief Title: The Effectiveness of Laser Acupuncture and Standard Medication Therapy on Mandibular Post-Odontectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Antonius Hapindra Kasim, doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-06-0952
Record Dates: First submitted 2023-08-27; First posted 2023-09-05 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Laser Acupuncture; Impacted Third Molar Tooth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Acupuncture and Standard Medication (Experimental): Laser Acupuncture: using RJ laser Nogier E program, with 4672Hz, 785 nm and power 70 mW. Dose 4 Joule at the acupuncture body points and 1 Joule at the ear points.
  Interventions: Device: Laser Acupuncture and Standard Medication
- Sham Laser Acupuncture and Standard Medication (Sham Comparator): Sham Laser Acupuncture: using RJ laser Nogier E program, with 4672Hz, 785 nm and power 70 mW. The laser is turned on but not activated
  Interventions: Device: Sham Laser Acupuncture and Standard Medication

INTERVENTIONS:
Device: Laser Acupuncture and Standard Medication — Laser Acupuncture: using RJ laser Nogier E program, with 4672Hz, 785 nm and power 70 mW. Dose 4 Joule at the acupuncture body points and 1 Joule at the ear points
  Arms: Laser Acupuncture and Standard Medication
Device: Sham Laser Acupuncture and Standard Medication — Laser Acupuncture: using RJ laser Nogier E program, with 4672Hz, 785 nm and power 70 mW. The laser is turned on but not activated
  Arms: Sham Laser Acupuncture and Standard Medication

SUMMARY:
Acute toothache is a problem that often occurs in the oral cavity. Toothache can be caused by an impacted tooth, in which the tooth cannot or will not erupt into its normal position. The American Association of Oral and Maxillofacial Surgeons (AAOMFS) states that 9 out of 10 people have at least one impacted tooth, and impacted mandibular third molars have the greatest prevalence. Laser acupuncture is an acupuncture modality that has the benefit of reducing pain after third molar extraction. The goal of this randomized controlled trial is to evaluate the group that received a combination of laser acupuncture and standard medication compared to the group that received the combination of sham laser acupuncture and standard medication alone, in management of post-mandibular odontectomy patients. The main objective of this study is to analyze the combination of laser acupuncture and medication significantly improving the patient's pain intensity, interincisal distance and post-odontectomy swelling compared to the combination group of sham laser acupuncture and medication.

DETAILED DESCRIPTION:
This is a clinical trial study to evaluate the group that received a combination of laser acupuncture and standard medication compared to the group that received the combination of sham laser acupuncture and standard medication alone, in management of post-mandibular odontectomy patients. The required sample was 57 mandibular third molars in male/female subjects post-odontectomy and randomized into 2 groups: (1) combination of laser acupuncture with standard medication and (2) combination of sham laser acupuncture with standard medication. The subjects will receive two times treatment, on day-1 (baseline) and day-3 after odontectomy. The outcome will be assessed on day-1 (baseline), day-3 and day-7 post-odontectomy. Patients and outcome assessors will be blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject
* Age 18 - 40 years
* Classification of Pell and Gregory class I, II and positions A, B, C
* Willing to participate in this research and sign informed consent

Exclusion Criteria:

* Pregnancy
* Have a history of using corticosteroid drugs in the last 3 months
* Have a history of medication with analgesics at least 24 hours before surgery
* Have an unstable systemic disease (such as uncontrolled hypertension and diabetes etc.)
* The patient has a medical emergency / hemodynamically unstable (such as having a hypertensive crisis)
* Wounds or skin diseases at the location of the acupuncture point irradiation
* Patients with a history of epilepsy
* High fever (> 38oC).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Day-1 (baseline), Day-3 and Day-7 post-odontectomy
  Rating scale for measuring pain, where the minimum value is 0 = no pain, and the maximum value is 100 = severe pain. A higher scale means worse outcomes.
Interincisal Space | Day-1 (baseline), Day-3 and Day-7 post-odontectomy
  Assess the maximum distance of opening the mouth (interincisal space) using calipers
Swelling | Day-1 (baseline), Day-3 and Day-7 post-odontectomy
  Assess the swelling dimensions using a tape measure

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia
Locations (1):
- Special dental and oral hospital, Faculty of Dentistry, University of Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes